CLINICAL TRIAL: NCT07330310
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Subcutaneous JKN2401 Injection in Patients With Moderate-to-Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Phase 3 Trial of JKN2401 Injection in COPD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Joincare Pharmaceutical Group Industry Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKN2401-III-01
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: JKN2401
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Injection, SC
  Interventions: Other: Placebo
- JKN2401 Injection (Experimental): JKN2401 Injection, SC dose A
  Interventions: Biological: JKN2401 Injection

INTERVENTIONS:
Biological: JKN2401 Injection — JKN2401 subcutaneous injection, Q4W
  Arms: JKN2401 Injection
Other: Placebo — Placebo subcutaneous injection,Q4W
  Arms: Placebo

SUMMARY:
A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Subcutaneous JKN2401 Injection in Patients With Moderate-to-Severe Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent; able and willing to comply with study procedures.
* Adults with documented COPD diagnosis and medical history consistent with guideline criteria.
* Relevant exposure history consistent with COPD (e.g., smoking and/or biomass exposure).
* On stable, guideline-based maintenance COPD therapy prior to randomization, per investigator judgment.
* Protocol-defined exacerbation history, symptom burden, and lung function at screening.

Exclusion Criteria:

* Current or past asthma, or other clinically significant respiratory disease that may confound assessment.
* Clinically significant uncontrolled comorbidities that increase risk or interfere with participation/outcomes.
* Immunodeficiency/immune dysregulation, active autoimmune disease requiring systemic immunosuppression, or significant opportunistic infection history.
* Active clinically significant infection or recent infection requiring systemic therapy; recent protocol-defined COPD exacerbation.
* Current/recent malignancy (except low-risk, adequately treated cancers per protocol) or clinically significant abnormal screening labs.
* Prohibited recent vaccines or therapies, prior relevant biologic/targeted therapy exposure, severe hypersensitivity to biologics/IMP, pregnancy/breastfeeding, or inability to comply (including substance abuse), per investigator judgment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of moderate or severe COPD exacerbations | during 52 weeks of treatment